CLINICAL TRIAL: NCT07035847
Title: Transcatheter Aortic Valve Replacement With Pure Echocardiography Guidance
Brief Title: TAVR With Echocardiography Guidance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Pan Xiangbin, Principle Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0501
Record Dates: First submitted 2025-05-11; First posted 2025-06-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Echo guided TAVR (Experimental): Patients received Echocardiography guided TAVR
  Interventions: Procedure: Echocardiography guided TAVR

INTERVENTIONS:
Procedure: Echocardiography guided TAVR — Echocardiography guided TAVR

SUMMARY:
This study aims to evaluate the safety and feasibility of performing transaxillary transcatheter aortic valve replacement (TA TAVR) guided solely by echocardiography in patients with severe aortic stenosis (AS).

ELIGIBILITY:
Inclusion Criteria:

1. symptomatic severe AS determined by echocardiography and Doppler that requiring aortic valve replacement, defined as: mean gradient ≥40 mmHg, peak aortic velocity ≥4 m/s, and aortic valve area (AVA) ≤1 cm2 (or an indexed AVA ≤0.6 cm2/m2)
2. a history of malignancy or a high familial risk of cancer, with refusal to undergo contrast- or radiation-guided procedures
3. chronic kidney disease and refuse to receive contrast agents or radiation exposure.
4. suitable for Transaxillary TAVR

Exclusion Criteria:

1. required hybrid procedures or concomitant interventions on other cardiac malformations
2. inoperable due to extremely high surgical risk or severe comorbidities
3. untreated clinically significant (>70% obstruction) proximal vessel coronary vascular disease amenable to revascularization
4. previously undergone aortic valve replacement.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Valve Academic Research Consortium-3 | 30 days after intervention
  Outcomes were reported according to the VARC-3 criteria.Which include: Technical success: Evaluated immediately post-procedure (e.g., successful vascular access, device delivery, deployment, no immediate complications).
  Device success: Includes successful valve function with acceptable hemodynamics and positioning.
  Procedural success: Includes 30-day outcomes, combining technical/device success and absence of major complications.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Pan, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided